CLINICAL TRIAL: NCT03336190
Title: Blue Star Cares: Innovative Approaches to Helping Military-Connected Caregivers
Acronym: BSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Blue Star Families (Unknown); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Wilcox Research (Unknown)
Responsible Party: Principal Investigator, Sherrie Wilcox, Principal Investigator, Uniformed Services University of the Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UP-17-00273
Record Dates: First submitted 2017-11-02; First posted 2017-11-08 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Military Family; Mental Health Disorder; Social Skills; Social Isolation; Communication; Quality of Life
Keywords: military; caregiver
MeSH Terms: conditions — Mental Disorders; Social Skills; Social Isolation; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Receives the full program, including the toolkit training and avatar interaction
  Interventions: Behavioral: avatar-based training

INTERVENTIONS:
Behavioral: avatar-based training — Interaction with an avatar-based module to practice skills learned during the toolkit training

SUMMARY:
The purpose of this project is to evaluate an interactive training program for military-connected caregivers (MCCs) of wounded warriors. The program leverages existing resources and incorporates evidence-based training and peer-based support networks to enhance continuity of care. The program consists of an educational Toolkit (workbook) and an avatar training interaction where an MCC can practice skills learned from the toolkit training with the avatar (how to navigate difficult conversations). This is an educational training evaluation to determine whether or not avatar interaction can effectively improve health outcomes in MCCs.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate an interactive training program for military-connected caregivers (MCCs) of wounded warriors. The program leverages existing resources and incorporates evidence-based training and peer-based support networks to enhance continuity of care. The program consists of an educational Toolkit (workbook) and an avatar training interaction where an MCC can practice skills learned from the toolkit training with the avatar (how to navigate difficult conversations). This is an educational training evaluation to determine whether or not avatar interaction can effectively improve health outcomes in MCCs.

The investigators will implement a pre-post design looking at a group of caregivers across multiple time points examining differences in outcomes from baseline (before engaging in the training/intervention) to after completing the training, including follow-ups at 3- and 6-months to evaluate longer-term outcomes.Those enrolled in the intervention will receive the complete training program (toolkit and avatar).

Project participants (i.e., MCCs who engage in the training and follow-up activities) will receive the (a) training toolkit workshop and will engage with the avatar to practice the knowledge and skills described in the workshop or will receive only the (b) training toolkit workshop (control).

Comparing the time differences will enable us to determine if the training program, specifically the avatar interaction, is associated with improved health and quality of life in caregivers of wounded warriors, enhanced caregiver social support and networks, improved patient (wounded warrior) experience of care, and reduced per capita costs of care for both the wounded warrior and caregiver.

Follow-up focus groups and interviews will be conducted to assess caregiver participant perspectives on what worked, what did not work, what they would like to see in the future, how the avatar interaction impacted them, and how the program could be improved in the future, as well as to clarify findings

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a military-connected caregiver over the age of 18.

Exclusion Criteria:

* Participants under the age of 18 or not a military-connected caregiver. Active duty military personnel are unable to participate in this project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life - Brief | Assess changes between baseline and 3 & 6 month follow-ups
  World Health Organization Quality of Life-Brief version (WHOQOL-BREF). The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials. The WHOQOL-BREF (Field Trial Version) produces a quality of life profile. It is possible to derive four domain scores. There are also two items that are examined separately: question 1 asks about an individual's overall perception of quality of life and question 2 asks about an individual's overall perception of their health. The four domain scores denote an individual's perception of quality of life in each particular domain. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score -
Social support | Assess changes between baseline and 3 & 6 month follow-ups
  Multidimensional Scale of Perceived Social Support, military version. Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS (Zimet et al., 1988) is a 12-item self-report measure that inquires about three dimensions of social relationships (family, friends, and a significant other) on a 7-point Likert-type scale (1 = very strongly disagree to 7 = very strongly agree). Higher scores on each of the subscales indicate higher levels of perceived support. A Global satisfaction with perceived support score can be obtained by taking the sum of the three scales. The current study added a fourth dimension relevant to military personnel that assessed sources of social support from military peers.
Depression | Assess changes between baseline and 3 & 6 month follow-ups
  Patient health questionnaire (PHQ)-2. Frequency of depressive symptoms were assessed with the 2-item Patient Health Questionnaire (PHQ-2). Items are rated on a 4-point scale from 0-3; higher scores indicate greater symptoms. Respondents then indicate the difficulty the symptoms have made their life on a 4 point scale, where high scores indicate greater difficulty.
Anxiety | Assess changes between baseline and 3 & 6 month follow-ups
  Generalized anxiety disorder-7.Frequency of anxiety symptoms were assessed using the 7-item Generalized Anxiety Disorder (GAD-7) (34). Items are rated on a 4-point scale, where 5, 10, and 15 are used as cutoffs for mild, moderate, and severe anxiety, respectively. Higher scores indicate greater symptoms
Caregiver somatic symptoms | Assess changes between baseline and 3 & 6 month follow-ups
  PATIENT HEALTH QUESTIONNAIRE (PHQ-15). For scoring, response options for these two symptoms are coded as 0 ("not at all"), 1 ("several days"), or 2 ("more than half the days" or "nearly every day"). Thus, the total PHQ-15 score ranges from 0 to 30 and scores of ≥5, ≥10, ≥15 represent mild, moderate and severe levels of somatization.

SECONDARY OUTCOMES:
Wounded warrior quality of life and health status | Assess changes between baseline and 3 & 6 month follow-ups
  World Health Organization Quality of Life-Brief version (WHOQOL-BREF). The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials. The WHOQOL-BREF (Field Trial Version) produces a quality of life profile. It is possible to derive four domain scores. There are also two items that are examined separately: question 1 asks about an individual's overall perception of quality of life and question 2 asks about an individual's overall perception of their health. The four domain scores denote an individual's perception of quality of life in each particular domain. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score -
Caregiver knowledge | Assess changes between baseline and 3 & 6 month follow-ups
  12 items assessing participant knowledge of caregiving. Items are rated on a 5-point scale where higher scores indicate higher knowledge of caregiving skills and responsibilities.
wounded warrior depression | Assess changes between baseline and 3 & 6 month follow-ups
  Patient health questionnaire (PHQ)-2. Frequency of depressive symptoms were assessed with the 2-item Patient Health Questionnaire (PHQ-2). Items are rated on a 4-point scale from 0-3; higher scores indicate greater symptoms. Respondents then indicate the difficulty the symptoms have made their life on a 4 point scale, where high scores indicate greater difficulty.
wounded warrior anxiety | Assess changes between baseline and 3 & 6 month follow-ups
  Generalized anxiety disorder-7.Frequency of anxiety symptoms were assessed using the 7-item Generalized Anxiety Disorder (GAD-7) (34). Items are rated on a 4-point scale, where 5, 10, and 15 are used as cutoffs for mild, moderate, and severe anxiety, respectively. Higher scores indicate greater symptoms
wounded warrior somatic symptoms | Assess changes between baseline and 3 & 6 month follow-ups
  PATIENT HEALTH QUESTIONNAIRE (PHQ-15). For scoring, response options for these two symptoms are coded as 0 ("not at all"), 1 ("several days"), or 2 ("more than half the days" or "nearly every day"). Thus, the total PHQ-15 score ranges from 0 to 30 and scores of ≥5, ≥10, ≥15 represent mild, moderate and severe levels of somatization.

OTHER OUTCOMES:
Costs of care | Assess changes between baseline and 3 & 6 month follow-ups
  Costs of care. Costs of care will be calculated based upon extent of injuries, frequency of visits, and projected annual costs based upon responses to outcomes across the study.
Common stressors | Assess changes between baseline and 3 & 6 month follow-ups
  Checklist of 14 common stressors. A checklist of 14 common stressors rated on a 10 point scale where higher scores indicate greater stress. Items included marital conflict, family conflict, and problems being a caregiver.
Relationship satisfaction and intimacy | Assess changes between baseline and 3 & 6 month follow-ups
  RELATIONSHIP ASSESSMENT SCALE. A 7-item scale designed to measure general relationship satisfaction. Respondents answer each item using a 5-point scale ranging from 1 (low satisfaction) to 5 (high satisfaction). Items 4 and 7 are reverse-scored. Scoring is kept continuous. The higher the score, the more satisfied the respondent is with his/her relationship.
medical outcomes | Assess changes between baseline and 3 & 6 month follow-ups
  12-Item Short Form Survey (SF-12). SF-12 measures physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. 2 items are used to estimate scores for four of the 8 health concepts (physical functioning: 0-5 where higher indicates more limited), role-physical: 0-3 where higher indicates more limited, role-emotional: 0-3 where higher indicates more limited, mental health: 0-11 where higher indicates more problems). Scores for the remaining 4 (bodily pain: 0-4 where higher indicates more problems, general health: 0-4 where higher indicates more problems, vitality, and social functioning: 0-4 where higher indicates more problems) are estimated using a single item each.
Wounded warrior satisfaction of care | Assess changes between baseline and 3 & 6 month follow-ups
  Patient Satisfaction Questionnaire 18 (PSQ-18). The short-form instrument, the PSQ-18, contains 18 items tapping each of the seven dimensions of satisfaction with medical care measured by the PSQ-III: general satisfaction (0-5, higher equals more disagreement), technical quality (0-5, higher equals more disagreement), interpersonal manner (0-5, higher equals more disagreement), communication (0-5, higher equals more disagreement), financial aspects (0-5, higher equals more disagreement), time spent with doctor (0-5, higher equals more disagreement), and accessibility and convenience (0-5, higher equals more disagreement). Items are rated on a 5 point scale where higher scores indicate more disagreement.
barriers to care | Assess changes between baseline and 3 & 6 month follow-ups
  15 item barriers to care survey. Respondents were asked about their use of professional physical or mental health services and about perceived barriers to physical and mental health treatment, particularly stigmatization as a result of receiving such treatment. Items are rated on a 2 point scale where higher scores indicate barriers. Overall scores range from 0-15 where higher scores indicate more barriers.
wounded warriors injury & pain | Assess changes between baseline and 3 & 6 month follow-ups
  Pain and injury checklist. Physical injuries were assessed with a 22-item checklist of body parts indicated on an image. Respondents could check locations of injuries. Number of injuries ranged from 0-22, where high scores indicate more injuries. Pain was rated on a 10-point scale where higher scores indicate more pain.
relationship happiness | Assess changes between baseline and 3 & 6 month follow-ups
  Relationship happiness with a single item, "Please slide the bar to the number, which best describes the degree of happiness, all things considered of your relationship" from 0-7 where higher scores indicate greater happiness.
Relationship quality | Assess changes between baseline and 3 & 6 month follow-ups
  Relationship quality with a single item, "We have a good marriage/partnership" rated on a 5 point scale where higher scores indicate greater happiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified data may be requested by emailing the Principal Investigator the specific research questions, variables of interest, analysis plan, and dissemination plan. Requests may be made at the completion of the study, once the main study questions have been evaluated and published.